CLINICAL TRIAL: NCT05727410
Title: A Phase II Trial of Neoadjuvant Nivolumab, Docetaxel, Cisplatin Therapy Followed by Surgery and Radiation Therapy for Resectable High Grade Salivary Gland Carcinoma
Brief Title: Neoadjuvant Nivolumab, Docetaxel, Cisplatin Therapy Followed by Surgery and Radiation Therapy for Resectable High Grade Salivary Gland Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Myung-Ju Ahn (Other)
Responsible Party: Sponsor-Investigator, Myung-Ju Ahn, M.D, Ph.D. Principal Investigator, Clinical Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-02-103
Record Dates: First submitted 2023-01-26; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: High-grade Salivary Gland Carcinoma
MeSH Terms: interventions — Nivolumab; Docetaxel

STUDY DESIGN:
Intervention Model Description: single-center trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nivolumab, docetaxel, cisplatin Group (Experimental): nivolumab, docetaxel, cisplatin (IV infusion every 3 weeks)
  Interventions: Drug: nivolumab, docetaxel, cisplatin Group

INTERVENTIONS:
Drug: nivolumab, docetaxel, cisplatin Group — Patients will be treated with nivolumab 360mg and plus docetaxel 60mg/m2 and cisplatin 60mg/m2 every 3 weeks for 3 cycles and will be evaluated for the operability. Patients with R0 resection will receive radiation 59.4 Gy in 27 fractions. Boost RT of 6.6 Gy in 3 fractions to tumor bed and/or gross tumor will be optional in patients who had R1-R2 resection. If tumors are regarded inoperable after neoadjuvant therapy (due to high risk of post-operative complication, or metastatic disease), they will be off from this study and receive the appropriate treatment, though they will be also included in the efficacy and safety analyses.

SUMMARY:
1. Primary Objective:

   - Major pathologic response rate defined by ≤ 10% of tumor composed of viable tumor
2. Secondary Objectives:

   * Complete resection rate
   * Response rate to neoadjuvant therapy according to RECIST 1.1
   * Downstaging at pathologic staging compared to clinical staging performed at study entry
   * Distant metastasis free survival (DMFS) rate at 2 years
   * Disease free survival at 2 years
   * Overall survival rate at 2 years
   * Safety and feasibility
3. Exploratory Objectives:

   * PD L1 expression by 28-8 immunohistochemistry
   * IHC (HER2, AR, etc)
   * Whole exome sequencing (WES)
   * Whole transcriptome sequencing (WTS)
   * Peripheral blood biomarkers (CD4+ T cells, CD8+ T cell, myeloid derived suppressor cells (MDSC), Treg etc)
   * Interferon gamma related gene expression profile
   * Multiplex florescence measure of tumor cells and tumor microenvironment cells

DETAILED DESCRIPTION:
This is a phase II, single center, open-label, single arm study in patients with resectable, high grade salivary gland carcinoma. Patients will be treated with nivolumab 360mg and plus docetaxel 60mg/m2 and cisplatin 60mg/m2 every 3 weeks for 3 cycles and will be evaluated for the operability. Patients with R0 resection will receive radiation 59.4 Gy in 27 fractions. Boost RT of 6.6 Gy in 3 fractions to tumor bed and/or gross tumor will be optional in patients who had R1-R2 resection. If tumors are regarded inoperable after neoadjuvant therapy (due to high risk of post-operative complication, or metastatic disease), they will be off from this study and receive the appropriate treatment, though they will be also included in the efficacy and safety analyses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically- or cytologically-confirmed resectable, clinically node-positive high grade salivary gland carcinoma Adenoid cystic carcinoma: Tubular/cribriform pattern predominant, Solid pattern > 30% Poorly differentiated carcinoma Mucoepidermoid carcinoma, High grade Polymorphous adenocarcinoma, High grade Lymphoepithelial carcinoma Salivary duct carcinoma Adenocarcinoma, NOS, High grade Carcinosarcoma Squamous cell carcinoma Carcinoma ex pleomorphic adenoma - risk is determined by type of carcinoma and extent of invasion
* No previous chemotherapy treatment history
* Patients who have at least 1 measurable or non-measurable lesion per the RECIST Guideline Ver. 1.1 as confirmed by imaging within 28 days before the first does of investigational product.
* Strongly encourage (but not must) to provide newly obtained core or excisional biopsy of a tumor lesion not previously treated.
* ECOG Performance Status Score 0 or 1
* Patients with a life expectancy of at least 3 months
* Patients whose latest laboratory data meet the below criteria within 28 days before the first dose of the investigational product. If the date of the laboratory tests at the time of enrollment is not within 28 days before the first dose of the investigational product, testing must be repeated within 28 days before the first dose of the investigational product, and these latest laboratory tests must meet the following criteria.

  * White blood cells ≥2,000/mm3 and neutrophils ≥1,500/mm3
  * Platelets ≥50,000/mm3
  * Hemoglobin ≥8.0 g/dL
  * AST (GOT) and ALT (GPT) ≤3.0-fold the upper limit of normal (ULN) of the study site
  * Total bilirubin ≤1.5-fold the ULN of the study site
  * Creatinine ≤1.5-fold the ULN of the study site or creatinine clearance (either the measured or estimated value using the Cockcroft-Gault equation) >45 mL/min
* Women of childbearing potential (including women with chemical menopause or no menstruation for other medical reasons) #1 must agree to use contraception#2 from the time of informed consent until 5 months or more after the last dose of the investigational product. Women must agree to use contraception#2 from the time of informed consent until 6 months or more after the last dose of docetaxel and 14 months or more after the last dose of cisplatin. Also, women must agree not to breastfeed from the time of informed consent until 5 months or more after the last dose of the investigational product. Women must agree not to breastfeed from the time of informed consent until 1 week or more after the last dose of docetaxel. Cisplatin has been reported to be found in human milk; women must agree not to breastfeed while receiving cisplatin.
* Men must agree to use contraception#2 from the start of study treatment until 7 months or more after the last dose of the investigational product, until 3 months or more after the last dose of docetaxel, and until 11 months or more after the last dose of cisplatin.

  * Women of childbearing potential are defined as all women after the onset of menstruation who are not postmenopausal and have not been surgically sterilized (e.g., hysterectomy, bilateral tubal ligation, bilateral oophorectomy). Postmenopause is defined as amenorrhea for ≥12 consecutive months without specific reasons. Women using oral contraceptives, intrauterine devices, or mechanical contraception such as contraceptive barriers are regarded as having childbearing potential.
  * The subject must consent to use any two of the following methods of contraception: vasectomy or condom for patients who are male or female subject's partner and tubal ligation, contraceptive diaphragm, intrauterine device, spermicide, or oral contraceptive for patients who are female or male subject's partner.

Exclusion Criteria:

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents except patient had no active treatment for past 5 years
* Patients who have received antineoplastic drugs (e.g., chemotherapy agents, molecular-targeted therapy agents, or immunotherapy agents) for high-grade SGC before the first dose of the investigational product
* Has received prior radiotherapy.
* Patients with residual adverse effects of prior therapy or effects of surgery that would affect the safety evaluation of the investigational product in the opinion of the investigator or sub-investigator.
* Patients with concurrent autoimmune disease or history of chronic or recurrent autoimmune disease
* Patients with any metastasis in the brain or meninx that is symptomatic or requires treatment.
* Patients with pericardial fluid, pleural effusion, or ascites requiring treatment
* Patients who have experienced a transient ischemic attack, cerebrovascular accident, or thrombosis within 180 days before enrollment
* Patients with a history of uncontrollable or significant cardiovascular disease meeting any of the following criteria:

  * Myocardial infarction within 180 days before enrollment
  * Uncontrollable angina pectoris within 180 days before enrollment
  * New York Heart Association (NYHA) Class III or IV congestive heart failure
  * Uncontrollable hypertension despite appropriate treatment (e.g., systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥ 90 mmHg lasting 24 hours or more)
  * Arrhythmia requiring treatment
* Patients with uncontrollable diabetes mellitus
* Patients with systemic infections requiring treatment
* Patients who have received systemic corticosteroids (except for temporary use, e.g., for examination or prophylaxis of allergic reactions) or immunosuppressants within 28 days before enrollment
* Patients who have undergone surgical adhesion of the pleura or pericardium within 28 days before enrollment
* Patients who have undergone surgery under general anesthesia within 28 days before enrollment
* Patients who have undergone surgery involving local or topical anesthesia within 14 days before enrollment
* Patients who have received any radiopharmaceuticals (except for examination or diagnostic use of radiopharmaceuticals) within 56 days before the first dose of the investigational product
* Women who are pregnant or breastfeeding, or possibly pregnant
* Patients who have received any other unapproved drug (e.g., investigational use of drugs, unapproved combined formulations, or unapproved dosage forms) within 28 days before enrollment
* Patients judged to be incapable of providing consent for reasons such as concurrent dementia
* Other patients judged by the investigator or sub-investigator to be inappropriate as subjects of this study
* Patient with current or past history of hypersensitivity to Nivolumab.
* Patients with current or past history of severe hypersensitivity to any other antibody products
* Patients with a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response rate defined by ≤ 10% of tumor composed of viable tumor | 6 months
  Primary tumors were assessed for the percentage of residual viable tumor that was identified on routine hematoxylin and eosin staining, and tumors with no more than 10% viable tumor cells were considered to have had a major pathological response. Patients who have progressive disease after neoadjuvant therapy and drop out from the study population will be counted as patients without major pathologic response.

SECONDARY OUTCOMES:
Complete resection rate | Up to 24 months
  Complete resection indicates a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed. Complete resection rate is defined as the percentage of the patients that underwent a resection and had a microscopically complete (or R0) resection.
Response rate to neoadjuvant therapy according to RECIST 1.1 | Up to 24 months
  RECIST 1.1 will be used as the primary measure for assessment of tumor response, date of disease progression, and as a basis for all protocol guidelines related to disease status (eg, discontinuation of study treatment).
Downstaging at pathologic staging compared to clinical staging performed at study entry | Up to 24 months
  Downstaging defined as pathologic TNM less than clinical TNM. Cancer staging calculator(AJCC 8th Edition)
Distant metastasis free survival (DMFS) rate at 2 years | Up to 24 months
  Distant metastases free survival (DMFS) is defined as the time between date of enrollment and the date of first diagnosis of distant metastasis or death, whichever comes first. Patients in whom distant metastases are discovered during neoadjuvant chemo/immunotherapy or the evaluation thereafter or at the immediate surgery, are considered to have an event at that time point.
Disease free survival at 2 years | Up to 24 months
  Patients that have undergone a resection and are alive without distant metastases (regardless of locoregional failure) are censored at the last date available.
Overall survival rate at 2 years | Up to 24 months
  Overall survival (OS) and is defined as the time between date of enrollment and date of death from any cause. Patients alive at last follow-up are censored at the last date available.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | Up to 24 months
  Who dose discontinued due to adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No